CLINICAL TRIAL: NCT04571203
Title: Phase I Study of Combined Deceased Donor Kidney and Hematopoietic Cell Transplants Using a Regimen to Promote Hematopoietic Cell Engraftment
Brief Title: Kidney and Hematopoietic Cell Transplants Using a Regimen to Promote Hematopoietic Cell Engraftment
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephan Busque, Professor of Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 57511
Record Dates: First submitted 2020-09-17; First posted 2020-09-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Immune Tolerance
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Intervention Model Description: End Stage Renal Disease subjects will receive a deceased donor kidney and vertebral body stem cell infusion. These transplant recipients post kidney transplant will undergo conditioning by ATG, Total Lymphoid irradiation and 1 single dose of TBI. Subsequently, the vertebral body stem cell infusion will be administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I Study of Combined DD Kidney and HCT Transplant (Experimental): Single arm Phase 1 non randomized dose finding study for safety, feasibility and efficacy of deceased donor vertebral body (VB) marrow cell infusion
  Interventions: Biological: Combined Deceased Donor Kidney and Hematopoietic Cell Transplants

INTERVENTIONS:
Biological: Combined Deceased Donor Kidney and Hematopoietic Cell Transplants — This combined kidney and hematopoietic cell transplants with a conditioning regimen with irradiation and ATG creates an environment of immune-tolerance. This promotes hematopoietic cell engraftment.
  Other Names: Radiation

SUMMARY:
This is a single arm phase 1 non randomized dose finding study for safety, feasibility and efficacy of deceased donor vertebral body (VB) marrow cell infusion and kidney transplantation.

DETAILED DESCRIPTION:
Patients will undergo a standard of care deceased donor kidney transplant and thereafter the recipient will receive TLI (Total Lymphoid Irradiation)/single low dose Total Body Irradiation, ATG (Anti-Thymocyte Globulin) conditioning, followed by an infusion of whole bone marrow cells harvested from the same donor vertebral bodies. Patients will be receive standard of care doses of steroids, MMF and tacrolimus as part of their transplant immunosuppression.

Subjects will be withdrawn from the immunosuppression if they have met the withdrawal criteria.

ELIGIBILITY:
Inclusion Criteria:

RECIPIENT INCLUSION CRITERIA:

1. Patient is ≥ 18 years old, and <65 years of age.
2. Has End Stage Renal Disease (ESRD) and is a de novo kidney transplant candidate part Stanford standard of care.
3. Listed with the Organ Procurement and Transplantation Network (OPTN) for deceased donor transplantation.
4. A serotypic (Human Leucocyte Antigen) HLA match with the donor of a least 1 locus in A, B or DR.
5. Males and females of reproductive potential who agree to practice a reliable form of contraception for at least 1 year post transplant.
6. Females have a negative serum pregnancy test.
7. Ability to understand and the willingness to sign a written informed consent document. Patients must have signed informed consent to participate in the trial.
8. No known contraindication to administration of rabbit ATG or low dose irradiation.

DONOR INCLUSION CRITERIA:

1. Brain dead donor aged ≥ 16 and ≤ 55
2. Organ Procurement Organization (OPO) consent for vertebral body procurement
3. Organ Procurement Organization consent for research
4. Projected cold ischemia time <24 hours.

Exclusion Criteria:

RECIPIENT EXCLUSION CRITERIA:

1. Known allergy to rabbit protein.
2. History of malignancy with the exception of non melanoma skin malignancy.
3. Pregnant woman or nursing mother.
4. Body weight >90kg or BMI >35.
5. Evidence of HIV 1/2 antibody (Ab), HTLV 1 and HTLV 2 Ab (Human T-Lymphotropic Virus), Hepatitis B sAg (surface antigen), Hepatitis C Ab, or positive syphilis screen.
6. EBV (Epstein Bar Virus)Ab positive donor to EBV Ab negative recipient.
7. Active bacterial, viral or fungal infection defined as currently taking medication for the infection.
8. Leukopenia (white blood cell count < 3000/mm3) or thrombocytopenia (with a platelet count < 100,000/mm3).
9. Psychiatric disorder(s) or psychosocial circumstance(s) which in the opinion of the Stanford Transplant team caring for this potential patient would place the patient at an unacceptable risk.
10. Concern for alcohol or other substance abuse.
11. Kidney disease at high risk for post transplant recurrence: aHUS (atypical hemolytic- uremic syndrome) and C3 glomerulopathy
12. Panel reactive antibody (PRA) >80%.
13. Positive donor specific antibody (DSA).
14. Prior or combined organ transplant.
15. Patients with >5 pack year smoking history, smoking within 10 years of enrollment, or first degree relative with lung cancer.

DONOR EXCLUSION CRITERIA:

1. History of malignancy with the exception of non melanoma skin malignancy.
2. History of autoimmune disease.
3. Known medical diagnosis of Zika virus infection within the prior 6 months, including post mortem screening.
4. Serological evidence of HIV, Hepatitis B (surface antigen positive), or Hepatitis C infection.
5. Evidence of systemic infection.
6. Kidney Donor Profile Index (KDPI) > 70%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients out of the total patients enrolled who received both the kidney and the bone marrow from the same donor. | 6 months
Determine the dose of TBI that will support donor CD3 Tcell chimerism between 30-75% at 45 days post infusion | day 45
  TBI dose in cGy associated with donor Tcell chimerism of >30 % immunosuppressive drug monotherapy.

SECONDARY OUTCOMES:
Number of patients who develop GVHD, all grades and types, within 60 months of kidney transplant | 60 months
Number of patients with either bacterial, viral or fungal infection within 12 months post transplant . | 12 months
Serum Creatinine | up to 60 months
Panel-Reactive Antibody (PRA) | Baseline, month 9, and month 12
  Report % of PRA on all participants
Donor-Specific Antibody (DSA) | Baseline, month 9, and month 12
  Report percentage of patients that develop DSA
Percentage of subjects on immunosuppressive medications after an eighteen month post transplant till month 60. | 60 months
Persistence of donor chimerism >1% | 3,6,9,12,15,18,24,48,60 months
  Percentage of patients with donor chimerism (any lineage)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, MD, Principal Investigator — Stanford University; Stephan Busque, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Busque S, Scandling JD, Lowsky R, Shizuru J, Jensen K, Waters J, Wu HH, Sheehan K, Shori A, Choi O, Pham T, Fernandez Vina MA, Hoppe R, Tamaresis J, Lavori P, Engleman EG, Meyer E, Strober S. Mixed chimerism and acceptance of kidney transplants after immunosuppressive drug withdrawal. Sci Transl Med. 2020 Jan 29;12(528):eaax8863. doi: 10.1126/scitranslmed.aax8863. PMID 31996467